CLINICAL TRIAL: NCT00226564
Title: The Effect of mu Opioid Receptor Polymorphism on the Response to Alfentanil During Lithotripsy
Brief Title: Genetic Determinants of Opioids Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yc19554-HMO-CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Alfentanil

INTERVENTIONS:
Drug: Alfentanil

SUMMARY:
The response to opioids varies greatly among individuals. Some of these variability is accounted for by genetic factors.

The present study was designed to evaluate the possibility that genetic polymorphism in the gene encoding for mu opioid receptor may explain variability in the response to alfentanil during lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20

Exclusion Criteria:

* Regular use of opioid drugs
* Known hypersensitivity to alfentanil

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1997-08

PRIMARY OUTCOMES:
Total alfentanil dose used during the procedure.
The extent of respiratory depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel